CLINICAL TRIAL: NCT02176629
Title: Usability of Virtual Reality in Subjects With Mild Cognitive Impairment or Alzheimer's Disease. MeMO-RV2
Brief Title: Usability of Virtual Reality in Subjects With Mild Cognitive Impairment or Alzheimer's Disease
Acronym: MeMO-RV2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 14-PP-03
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: MCI; Alzheimer's Disease
Keywords: Virtual Reality; mild cognitive impairment; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Condition virtual reality (VR) (Experimental): The subject is placed in front of a Barcotm screen capable of displaying high quality images.
  Interventions: Other: Condition virtual reality (VR) then Condition classic cognitive stimulation (CCS)
- Condition classic cognitive stimulation (CSC) (Active Comparator): It is proposed about using the test dam Zazzo suitable for elderly. This classic test measures sustained attention.
  Interventions: Other: Condition classic cognitive stimulation (CCS) then Condition virtual reality (VR)

INTERVENTIONS:
Other: Condition virtual reality (VR) then Condition classic cognitive stimulation (CCS)
  Arms: Condition virtual reality (VR)
Other: Condition classic cognitive stimulation (CCS) then Condition virtual reality (VR)
  Arms: Condition classic cognitive stimulation (CSC)

SUMMARY:
Cognitive and memory problems characterize Alzheimer's disease (AD). Along with these disorders, psychological and behavioral symptoms (also known as neuropsychiatric symptoms) , as well as pathophysiological processes are frequently found and involved significantly in maintaining autonomy, prognosis and treatment of the disease. Apathy or disorder motivation is the most common disorder behavior and early stages of cognitive impairment. Apathy is particularly associated with cognitive difficulties such as attention deficit disorder - concentration.

In terms of prevention as term care , there is now a broad consensus that interventions on cognition and behavior must not be limited to pharmacological treatment but should also promote non-drug approaches.

Interest in video games (serious games and serious games) as intervention support rehabilitation is growing. Similarly, the virtual reality (VR) and the new information technologies and communications offer significant opportunities in terms of rehabilitation and therapeutic assistance.

This protocol is part of a European project to propose techniques for improving the treatment of people at risk of social exclusion ( VERVE project ) aims .

A first experiment conducted in 2013 showed the acceptability of Virtual Reality (VR) in healthy elderly subjects. In a second step , it is important to validate the feasibility of using the RV or in frail subjects with mild cognitive impairment or Alzheimer's disease in mild to moderate in a clinical environment.

This is a biomedical , randomized given to a group of patients with mild cognitive impairment or Alzheimer's disease & diseases associated with mild to moderate.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 60 years.
* Introducing either:

  * MCI diagnosis (ICD-10)
  * diagnosis of Alzheimer's disease or mixed mild to moderate (ICD 10).
* Subject undisturbed locomotion requiring the use of a walking aid.
* Score at the Mini Mental Test (MMSE) between 16 and 28.

Exclusion Criteria:

* Presence of psychiatric disorders
* Presence of eye diseases causing blurred vision can not be corrected with lenses or glasses.
* Presence of auditory pathologies causing a significant decrease in hearing unaided.
* High sensitivity to motion sickness.
* migraine disease.
* Subject epileptic.
* Subject vulnerable

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Evaluate the acceptability of the RV | At the end of experience (45 min)
  Analog scale assessment of satisfaction from 0 to 100% is given at the end of experience about that evaluates:
  * The general acceptability of the RV
  * His sense of security
  * The environment of RV
  * The degree of motivation

SECONDARY OUTCOMES:
Evaluate the motivation of subjects (interest, cognition) is greater in the virtual environment during the VR experience compared to a conventional cognitive stimulation activity (CSC). | At the end of experience (45 min)
  * Percentage of membership: relationship between time spent playing in the subject and the total time required by the experiment (Comparison of the two conditions (RV vs SCC));
  * Degree of performance: number of "cognitive targets" found by the subject during the experiment. (Comparison of the two conditions (RV vs SCC));
  * Degree of attention: the number of errors in target detection;
  * Evaluation of the degree of presence of participants (condition RV) using the ITC-SOPI.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ROBERT, PUPH, Study Director — Centre Hospitalier Universitaire de Nice
Locations (1):
- Institut Claude Pompidou, Nice, France